CLINICAL TRIAL: NCT00742482
Title: A Phase III Study With Freeze Dried HL10, Three Dosages of 200 mg/kg Ideal Body Weight Versus Standard Therapy in ALI/ARDS Patients
Brief Title: Efficacy and Safety of 3 Doses of HL10 Given at Fixed Time Intervals Compared to Standard Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A 300 patient safety analysis by the Data Monitoring Committee showed a trend towards higher mortality in the treatment group.
Sponsor: LEO Pharma (Industry)
Responsible Party: Edmée Steenken/Project Co-ordinator, LEO Pharma A/S
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL 0101 INT
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2009-02

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: HL 10 — Freeze dried HL 10

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of three doses of HL 10 given at fixed time intervals compared to standard therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients intubated and on mechanical ventilation
* Patients with Acute Lung Injury defined as (a, b, c and d are all applicable): a: PaO2/FiO2 < or equal to 300 mmHg (40.0 kPa) (regardless of PEEP level), b: Acute onset, c: Pulmonary artery wedge pressure < or equal to 18 mmHg when measured or no clinical evidence of left atrial hypertension, d: Bilateral infiltrates seen on frontal chest radiograph
* Less than 60 hours from onset of the present period of mechanical ventilation to 1st instillation
* Expected to continue on mechanical ventilation for more than 24 hours
* 18 years of age or older
* Following receipt of verbal and written information about the trial, the patient or legally acceptable representative must provide signed and dated informed consent before any trial related activity is carried out

Exclusion Criteria:

* Current diagnosis of acute bronchial asthma attack
* History of or clinical suspicion of lung fibrosis
* Current diagnosis of suspected pulmonary thrombo-embolism
* Patients on daily medication for chronic obstructive pulmonary disease at time of admission to ICU
* Patients who have received mechanical ventilation for more than 48 hours continuously within 1 month prior to the present period of mechanical ventilation
* Patients with pneumonectomy or lobectomy
* Patients with untreated pneumothorax at time of instillation
* Patients having tracheostomy at time of instillation
* Patients who have had surgical procedures under general anaesthesia performed within 6 hours prior to inclusion blood gas sample
* Patients having mean arterial blood pressure < 50 mmHg in spite of adequate fluid administration and/or vasoactive drugs at time of instillation
* Patients having PaO2 < 75 mmHg with a FiO2 = 1.0 not responding to adjustment of PEEP at time of instillation
* Glasgow Coma Score < or equal to 10 before sedation or major findings on CT/MR scan of the head such as: brain oedema, acute space occupying lesion, other acute lesions with bleeding or mass effect (patients with minor lesion which do not require further diagnostics or monitoring can be included)
* Patients with life expectancy less than 3 months due to primary disease assessed by the attending physician (e.g., end-stage cancer, AIDS or generally poor health)
* Known or suspected hypersensitivity to constituents(s) of the investigational product
* Patients who have received treatment with any investigational drug within the previous 4 weeks
* Current participation in any other interventional clinical trial until day 29 of the trial
* Patients previously randomised in this trial
* Patients known or suspected of not being able to comply with a study protocol (e.g., due to alcoholism, drug dependency or psychotic state)
* Females of childbearing potential who have a positive pregnancy test or who are breast feeding
* Patients suffering from highly infectious diseases where trial related procedures could pose a safety risk for the staff (e.g., SARS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
28 days mortality | 28 days

SECONDARY OUTCOMES:
Days alive and off ventilator | Day 29
Days on ventilation | Day 1 to Day 29
Days alive and out of ICU | Day 29
Changes in Pao2/FiO2 ratios and other relevant lung parameters, changes in SOFA score | From Day 1 to Day 4, Day 1 to Day 8, Day 4 to Day 8
Dead/alive at discharge of ICU | Followed until Day 180
Dear/alive at discharge from hospital | Followed until Day 180
180 days mortality | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Kesecioglu, MD, PhD, Principal Investigator — Anaesthesist-Intensivist, Department of Intensive Care Medicine
Locations (13):
- Allgemeines Krankenhaus, Klinik für Anästhesie un Allgemeine Intensivmedizin, Vienna, Austria
- Erasme University Hospital, Brussels, Belgium
- Mount Sinai Hospital, Critical Care Unit, Toronto, Ontario, Canada
- Odense University Hospital, Odense C, Denmark
- Kuopio University Hospital, Intensive Care Unit, Kuopio, Finland
- Hôpital Pitié Salpétrière, Département d'Anesthésie Réanimation, Paris, France
- Klinik für Anästhesiologie der RWTH Aachen, Aachen, Germany
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - Department of Intensive Care Medicine, Utrecht
- Ullevål University Hospital, INtensive Care Department, Oslo, Norway
- Consorci Hospitalari Parc Taulí, Sabadell (Barcelona), Spain
- University Hospital of Lund, Department of Intensive Care, Lund, Sweden
- St Thomas Hospital, Adult Intensive Care, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu Q, Zhang M, Girardi C, Bouhemad B, Kesecioglu J, Rouby JJ. Computed tomography assessment of exogenous surfactant-induced lung reaeration in patients with acute lung injury. Crit Care. 2010;14(4):R135. doi: 10.1186/cc9186. Epub 2010 Jul 15. PMID 20633284
- [Derived] Kesecioglu J, Beale R, Stewart TE, Findlay GP, Rouby JJ, Holzapfel L, Bruins P, Steenken EJ, Jeppesen OK, Lachmann B. Exogenous natural surfactant for treatment of acute lung injury and the acute respiratory distress syndrome. Am J Respir Crit Care Med. 2009 Nov 15;180(10):989-94. doi: 10.1164/rccm.200812-1955OC. Epub 2009 Aug 27. PMID 19713451